CLINICAL TRIAL: NCT02842151
Title: Optimizing the Assessment of Refractive Outcomes After Cataract Surgery and Implantation of a Monofocal IOL
Brief Title: Optimizing the Assessment of Refractive Outcomes After Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: ILQ732-I001
Record Dates: First submitted 2016-07-14; First posted 2016-07-22 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-11

CONDITIONS: Cataract
Keywords: Intraocular Lens (IOL)
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Manifest refraction (Other): Manifest refraction performed by autorefraction (automated) and manual procedures (standard). Subject implanted with ACRYSOF® IQ Monofocal IOL Model SN60WF. Autorefraction performed by Topcon® KR-1W Wave-Front Analyzer.
  Interventions: Procedure: Manifest refraction; Device: ACRYSOF® IQ Monofocal IOL Model SN60WF; Device: Topcon® KR-1W Wave-Front Analyzer

INTERVENTIONS:
Procedure: Manifest refraction — Manifest refraction performed by autorefraction (automated) and manual procedures (standard)
Device: ACRYSOF® IQ Monofocal IOL Model SN60WF — Monofocal IOL implanted for long-term use over the lifetime of the cataract patient
Device: Topcon® KR-1W Wave-Front Analyzer — Wavefront and topography system used to obtain autorefraction data

SUMMARY:
The purpose of this study is to evaluate current available assessments (automated vs. manual) with which manifest refraction data and biometric variables are obtained to understand if data from an automated refractor can be utilized to optimize the A-constant as well as manual subjective refraction (ie, to a clinically insignificant difference). The A-constant is the calculated number that helps the surgeon determine which IOL should be implanted in the eye during cataract surgery.

DETAILED DESCRIPTION:
Subjects will be implanted with ACRYSOF® IQ Monofocal IOL Model SN60WF. Standard clinical practice will be followed for pre-operative testing, IOL power estimation and IOL implantation. Only one eye will be enrolled in the study per surgeon determination. The eye will undergo both an automated and manual manifest refraction assessment at 3 months postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an Ethics Committee/Institutional Review Board approved Informed Consent;
* Willing and able to attend all scheduled study visits as required per protocol;
* Diagnosed with cataract in one or both eyes;
* Planned cataract removal by phacoemulsification with implantation of a monofocal IOL; laser refractive procedures for incisions (primary and sideport), capsulorhexis and lens fragmentation are allowed;
* Preoperative keratometric astigmatism ≤ 1.0 diopter (D);
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential, pregnant, or breast-feeding;
* History of ocular pathology, ocular inflammation, or ocular conditions, as specified in the protocol;
* Previous intraocular or corneal surgery;
* Use of systemic medications that, in the opinion of the Investigator, may confound the outcome or increase the risk of complications to the subject;
* Any medical condition that, in the opinion of the Investigator, may confound the results of this study, prohibit the completion of the study assessments, or increase the risk for the subject;
* Other protocol-defined exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, A Novartis Division, Study Director — Alcon, A Novartis Division

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 investigative sites located in Ireland (1) and the US (2).
Pre-assignment Details: Of the 162 enrolled, 12 subjects were exited as screen failures prior to intraocular lens (IOL) implantation. This reporting group includes all subjects with attempted implantation (150).
Groups:
- Overall: Subjects implanted with ACRYSOF® IQ Monofocal IOL Model SN60WF.
Period: Overall Study
Arm/Group | Overall
Started (All subjects with attempted implantation (successful or aborted) (Safety Analysis Set)) | 150
Completed | 148
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Subject moved too far away | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all eyes with successful IOL implantation (All-Implanted Analysis Set).
Arm/Group | Overall
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 131
  Unknown or Not Reported | 16

OUTCOME MEASURES:

1. Primary Outcome: IOL A-constant at 3 Months at Each Site
Description: The A-constant, is a type of IOL constant, that accounts for clinical variables that may affect the refractive outcome (e.g. patient factors, biometry method). It relates the power of the IOL to axial length and corneal measurements. It is specific to the design of the IOL, style, and placement within the eye. The optimization of the A-constant is fundamental to achieving the targeted refractive outcomes, offset any observed error and for ensuring high patient satisfaction following cataract surgery. Since errors/noise from refraction plays a significant role in A-constant optimization, it is important to determine if an automated method has any advantages over conventional manifest refraction. A-constants based on autorefraction and manifest refraction for the study eye are compared for each subject. The mean difference between the two methods cannot be greater than 0.15 D at each of the three study centers for the methods to be considered equivalent.
Time Frame: Month 3 (Day 80-100) Post Study Eye Implantation
Population: All-Implanted Analysis Set with non-missing data
Measure: Mean (Standard Deviation); unit: unitless
Units Other Than Participants: Eyes
Groups:
- Manifest Refraction: Standard manifest refraction assessed with an ETDRS chart using a phoropter
- Autorefraction: Autorefraction performed by Topcon® KR-1W Wave-Front Analyzer
Arm/Group | Manifest Refraction | Autorefraction
Number analyzed (Participants) | 147 | 147
Number analyzed (Eyes) | 147 | 147
unitless
  Study Site 1 (US): number analyzed (Participants) | 52 | 52
  Study Site 1 (US): number analyzed (Eyes) | 52 | 52
  Study Site 1 (US) | 119.23 (0.408) | 119.18 (0.493)
  Study Site 2 (US): number analyzed (Participants) | 53 | 53
  Study Site 2 (US): number analyzed (Eyes) | 53 | 53
  Study Site 2 (US) | 118.86 (0.601) | 118.93 (0.723)
  Study Site 3 (Ireland): number analyzed (Participants) | 42 | 42
  Study Site 3 (Ireland): number analyzed (Eyes) | 42 | 42
  Study Site 3 (Ireland) | 118.39 (3.071) | 118.52 (3.137)
Statistical Analysis 1: Comparison: Manifest Refraction vs Autorefraction; To demonstrate equivalency at Site 1, A-constant with manifest refraction was compared to A-constant with autorefraction; Test type: Equivalence — Difference in A-Constant is manifest refraction minus autorefraction. The criteria for equivalence (based on paired difference t-test) was established if the bounds of the 90% two-sided confidence interval (CI) on the difference was contained within the equivalence range (-0.15, 0.15); Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-0.03 to 0.13], Standard Deviation 0.346
Statistical Analysis 2: Comparison: Manifest Refraction vs Autorefraction; To demonstrate equivalency at Site 2, A-constant with manifest refraction was compared to A-constant with autorefraction; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.07, 90% CI 2-sided [-0.21 to 0.07], Standard Deviation 0.595
Statistical Analysis 3: Comparison: Manifest Refraction vs Autorefraction; To demonstrate equivalency at Site 3, A-constant with manifest refraction was compared to A-constant with autorefraction; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.13, 90% CI 2-sided [-0.22 to -0.04], Standard Deviation 0.340

ADVERSE EVENTS:
Time Frame: IOL implantation through study completion, an average of 3 months
Description: Adverse Events (AEs) were defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the clinical investigation. Safety Analysis Set
Groups:
- Ocular Adverse Events: At risk population for ocular adverse events is included with units of eyes.
- Non-ocular Adverse Events: At risk population for non-ocular adverse events is included with units of subjects.
Arm/Group | Ocular Adverse Events | Non-ocular Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 4/150 | 2/150
Other Adverse Events (participants affected / at risk) | 9/150 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ocular Adverse Events (N=150) | Non-ocular Adverse Events (N=150)
Intraocular pressure increased (Investigations) | 3 | 0
Cystoid macular oedema (Eye disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ocular Adverse Events (N=150) | Non-ocular Adverse Events (N=150)
Eye inflammation (Eye disorders) | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02842151/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT02842151/SAP_001.pdf